CLINICAL TRIAL: NCT02925026
Title: Lactoferrin and Lysozyme Supplementation for Environmental Enteric Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Malawi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lactoferrin-Lysozyme
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Environmental Enteric Dysfunction
MeSH Terms: interventions — Lactoferrin; Muramidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactoferrin+Lysozyme (Experimental): lactoferrin and lysozyme in rice flour
  Interventions: Dietary Supplement: Lactoferrin; Dietary Supplement: Lysozyme
- Placebo (Placebo Comparator): rice flour
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactoferrin
  Arms: Lactoferrin+Lysozyme
Dietary Supplement: Lysozyme
  Arms: Lactoferrin+Lysozyme
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo controlled trial of daily lactoferrin and lysozyme supplementation in improving environmental enteric dysfunction in Malawian children

ELIGIBILITY:
Inclusion Criteria:

* children aged 12-35 months
* youngest eligible child in each household

Exclusion Criteria:

* severe or moderate acute malnutrition
* severe chronic illness
* children unable to drink 20 mL of dual sugar solution
* children in need of acute medical treatment for illness or injury at time of enrollment

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Dual Sugar Absorption Test | 8 weeks
  lactulose-mannitol ratio in urine
Dual Sugar Absorption Test | 16 weeks
  lactulose-mannitol ratio in urine

SECONDARY OUTCOMES:
Lactulose Excretion | 8 weeks
  percentage of ingested lactulose excreted in urine
Lactulose Excretion | 16 weeks
  percentage of ingested lactulose excreted in urine
Mannitol Excretion | 8 weeks
  percentage of ingested mannitol excreted in urine
Mannitol Excretion | 16 weeks
  percentage of ingested mannitol excreted in urine

OTHER OUTCOMES:
Linear Growth | 16 weeks
  changes in linear growth

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Principal Investigator — Washington University in St. Louis; University of Malawi; Chrissie Thakwalakwa, PhD, Study Director — Study Director; Indi Trehan, MD MPH DTM&H, Study Director — Washington University in St. Louis; University of Malawi
Locations (1):
- Malawi, Blantyre, Malawi

REFERENCES:
- [Derived] Cheng WD, Wold KJ, Benzoni NS, Thakwalakwa C, Maleta KM, Manary MJ, Trehan I. Lactoferrin and lysozyme to reduce environmental enteric dysfunction and stunting in Malawian children: study protocol for a randomized controlled trial. Trials. 2017 Nov 6;18(1):523. doi: 10.1186/s13063-017-2278-8. PMID 29110675